CLINICAL TRIAL: NCT00201006
Title: Treatment of Obesity in Underserved Rural Settings (TOURS)
Acronym: TOURS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 273; R01HL073326 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2014-03-07 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Face-to-face counseling (Experimental): 26 biweekly face-to-face group counseling sessions
  Interventions: Behavioral: Face-to-face counseling
- Telephone Counseling (Experimental): 26 biweekly telephone counseling sessions
  Interventions: Behavioral: Telephone counseling
- Mail contact (Active Comparator): 26 biweekly newsletters with weight management advice
  Interventions: Other: Mail contact

INTERVENTIONS:
Behavioral: Face-to-face counseling — Biweekly group behavioral counseling sessions conducted in a face-to-face format
  Arms: Face-to-face counseling
Behavioral: Telephone counseling — Biweekly telephone counseling sessions conducted in a one-on-one format
  Arms: Telephone Counseling
Other: Mail contact — Biweekly written newsletters with weight management advice delivered via U.S. mail
  Arms: Mail contact

SUMMARY:
To test the effectiveness of interventions designed to promote long-term weight management of obese women in medically underserved rural counties.

DETAILED DESCRIPTION:
BACKGROUND:

The recent dramatic rise in the prevalence of obesity has heightened awareness of the significant impact of overweight, physical inactivity, and unhealthy eating patterns on the development of chronic diseases and disability While there is little doubt that obesity and associated lifestyle factors (e.g., sedentary lifestyle) constitute serious threats to health, it is also clear that lifestyle interventions can produce body weight reductions of sufficient magnitude to improve health. The existing research is limited, however, with respect to two important factors, specifically, its generalizability to underserved populations, and the maintenance of treatment effects. Most weight-loss trials have consisted of efficacy studies conducted with middle-class participants and delivered in "optimal" (i.e., academic research) venues rather than in "real world" (i.e., community) settings. Furthermore, the existing literature shows that, in the absence of long-term care, a regaining of lost weight routinely follows the conclusion of treatment. Recent research has shown improved maintenance of lost weight when lifestyle interventions are supplemented with clinic-based follow-up programs. Thus, the next logical steps in this line of research are (a) to extend these studies to community settings with underserved populations and (b) to test promising alternative and potentially more efficient modes of treatment delivery, such as follow-up care via telephone-based contacts rather than via in-person clinic visits.

DESIGN NARRATIVE:

A randomized controlled clinical trial will examine the impact of two maintenance interventions designed to sustain weight lost in lifestyle treatment of obesity. The study sample will include 300 obese women, ages 50-75 years, from medically underserved rural areas in North Central Florida. All participants will receive a 6-month lifestyle intervention for weight loss (called Phase 1) followed by randomization to one of three 12-month follow-up (called Phase 2) programs: (A) a Face-to-Face Office-Based Maintenance Program, (B) a Telephone-Based Maintenance Program, or (C) an Education Comparison Condition. Participants will be stratified according to county and to BMI, and randomly assigned in groups of 11-12 to one of the two experimental programs or to the comparison condition. The experimental maintenance programs are designed to help participants sustain the eating and physical activity patterns needed to maintain lost weight. The primary difference between the two maintenance programs is their mode of delivery. One will be delivered via an office-based group counseling format; the other will be delivered via telephone counseling. The education comparison condition will involve a program of print materials on the maintenance of a healthy lifestyle delivered via biweekly newsletters.

ELIGIBILITY:
Inclusion criteria:

BMI between 30 and 45

Exclusion criteria:

presence of serious disease

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2003-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Perri, PhD, Principal Investigator — University of Florida

REFERENCES:
- [Result] Perri MG, Limacher MC, Durning PE, Janicke DM, Lutes LD, Bobroff LB, Dale MS, Daniels MJ, Radcliff TA, Martin AD. Extended-care programs for weight management in rural communities: the treatment of obesity in underserved rural settings (TOURS) randomized trial. Arch Intern Med. 2008 Nov 24;168(21):2347-54. doi: 10.1001/archinte.168.21.2347. PMID 19029500

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study announcements were mailed to households in 6 rural counties in northern Florida designated in whole or in part as health professional shortage areas. Women who responded to the announcements were invited to an orientation/screening session wherein informed consent was obtained. Height and weight were measured by a registered nurse.
Pre-assignment Details: 298 women participated in a standard 6-month lifestyle modification program for weight loss, delivered in groups at Cooperative Extension Offices. Eligibility for randomization required completion of the 6-month lifestyle program; 234 completed the initial treatment and were assigned randomly to one of the three extended care conditions.
Period: Overall Study
Arm/Group | Face-to-face Counseling | Telephone Counseling | Mail Contact
Started | 83 | 72 | 79
Completed | 75 | 70 | 75
Not Completed | 8 | 2 | 4
Not completed — Withdrawal by Subject | 7 | 2 | 3
Not completed — Adverse Event | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Face-to-face Counseling | Telephone Counseling | Mail Contact | Total
Number analyzed (Participants) | 83 | 72 | 79 | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (6.2) | 59.8 (6.2) | 58.6 (6.0) | 59.4 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 72 | 79 | 234
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 83 | 72 | 79 | 234
Body weight [Mean (Standard Deviation); unit: kg] | 97.8 (14.3) | 96.4 (16.8) | 95.0 (13.4) | 96.4 (15.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight.
Description: Change in body weight during the 12-month period following completion of a 6-month lifestyle treatment for obesity.
Time Frame: one year
Population: Data from all randomized participants were analyzed according to the Intent to Treatment principle. Missing data (6%) were completed based on known pattern of weight regain (i.e., 0.3 kg per month).
Measure: Mean (Standard Error); unit: kg
Arm/Group | Face-to-face Counseling | Telephone Counseling | Mail Contact
Number analyzed (Participants) | 83 | 72 | 79
kg | 1.2 (0.6) | 1.2 (0.7) | 3.7 (0.7)

ADVERSE EVENTS:
Time Frame: 1 year
Description: self-reporting by participants
Groups:
- Face-to-face: received 26 biweekly office-based, face-to-face group counseling sessions
- Telephone: received 26 biweekly individual telephone counseling sessions
- Mail: received by mail 26 biweekly newsletters with weight management information
Arm/Group | Face-to-face | Telephone | Mail
Serious Adverse Events (participants affected / at risk) | 21/83 | 20/72 | 12/79
Other Adverse Events (participants affected / at risk) | 19/83 | 9/72 | 12/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Face-to-face (N=83) | Telephone (N=72) | Mail (N=79)
cardiac symptom (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
circulatory problems (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
ear problems (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
eye problem (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
gynecologic and breast problems (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 2 (2)
kidney problem (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
musculoskeletal injury (Musculoskeletal and connective tissue disorders) | 14 (14) | 11 (11) | 6 (6)
neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
neurological symptoms (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
respiratory problem (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
thyroid problem (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Face-to-face (N=83) | Telephone (N=72) | Mail (N=79)
minor musculoskeletal injuries (Musculoskeletal and connective tissue disorders) | 19 (19) | 9 (9) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No